CLINICAL TRIAL: NCT01059279
Title: Heat Intolerance in the Group of FMF Patients
Status: Terminated | Type: Observational
Why Stopped: unable to recruit patients
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof.Avi Livneh, Professor, Sheba Medical Center
Other Study IDs: SHEBA-09-7575-AL-CTIL
Record Dates: First submitted 2010-01-28; First posted 2010-01-29 (Estimated); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Familial Mediterranean Fever; Heat Intolerance; Heat Tolerance Test
Keywords: Familial Mediterranean fever; Cytokines; Inflammatory proteins; MEFV; mutations; Heat Intolerance; Heat Tolerance Test
MeSH Terms: conditions — Familial Mediterranean Fever

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- FMF patients: 15 FMF patients with double mutations MEFV, mail sex, from the age from 18 to 30. treated with colchicine, without attacks not less than 2 months
- healthy people: Healthy individuals, that participated in the study of Heller Institute of Medical Research.

SUMMARY:
There now causation between Heat Intolerance and FMF that were showed in studies till now. We suggest that the prevalence of Heat Intolerance in the group of the FMF patients will be significantly higher than in the group of healthy individuals, that participated in the study of Heller Institute of Medical Research. The aim of the study is verification of causation between these pathologies. The information obtained by the study may allow us to determine the sequence of events associated with FMF attack development, and perhaps take us one step further in the understanding of the pathogenesis of the disease.

15 FMF patients with double mutations MEFV, mail sex, from the age from 18 to 30 without attacks during not less than 2 month will participate in the study. To identify an individuals susceptibility to exercise heat test, a Heat Tolerance Test (HTT) will perform, according to HTT Protocol of Heller Institute of Medical Research.

DETAILED DESCRIPTION:
Familial Mediterranean fever (FMF) is a genetic disease, caused by mutations in the FMF gene, entitled MEFV. The disease is characterized by painful attacks of inflammation in sites lined by serous membranes (e.g. abdominal pain caused by inflammation of the peritoneum, a serous membrane surrounding all internal organs within the abdomen, fever during the attack. Continuous colchicine treatment prevents attacks in most patients. The pathogenesis of the disease, what leads to the attacks, is the questions not yet resolved. We know that there is correlation between protein Pyrin and activity of Interleukin 1 (IL1).

Tolerance to sustain heat stress varies due to individual variation. Under extreme conditions of exercise-heat stress, even healthy, well acclimated, physically fit individuals will ultimately store heat at the rate that will cause body temperature to rise. Individuals who are not able to sustain heat and whose body temperature will start rising earlier and at a higher rate than that of others, under the same conditions, are defined as "heat intolerant".

There now causation between Heat Intolerance and FMF that were showed in studies till now. We suggest that the prevalence of Heat Intolerance in the group of the FMF patients will be significantly higher than in the group of healthy individuals, that participated in the study of Heller Institute of Medical Research. The aim of the study is verification of causation between these pathologies. The information obtained by the study may allow us to determine the sequence of events associated with FMF attack development, and perhaps take us one step further in the understanding of the pathogenesis of the disease.

15 FMF patients with double mutations MEFV, male sex, from the age from 18 to 30 without attacks during not less than 2 month will participate in the study. To identify an individuals susceptibility to exercise heat test, a Heat Tolerance Test (HTT) will perform, according to HTT Protocol of Heller Institute of Medical Research.

ELIGIBILITY:
Inclusion Criteria:

* double mutations MEFV
* mail
* age from 18 to 30
* colchicine treatment
* absence of attack during 2 months

Exclusion Criteria:

* individual wish

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: 15 FMF patients with double mutations MEFV, mail sex, from the age from 18 to 30. treated with colchicine, without attacks not less than 2 months
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2009-12; Primary Completion 2012-08 (Actual); Study Completion 2024-03-03 (Actual)

PRIMARY OUTCOMES:
Rate of heat intolerance defined by the HTT protocol of Heller Institute of Medical Research. | At the end of the test - One day test
  Number of patients who failed the HTT divided by number of patients undergoing the test. Failure to finished the test for reasons other than a rise in the temperature will be excluded

CONTACTS AND LOCATIONS:
Overall Officials: Avi Livneh, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel